CLINICAL TRIAL: NCT06315283
Title: A 21-Week, Multicenter, Open-Label, Multiple-Dose Trial to Assess the Comparative Bioavailability of Olanzapine Prolonged-Release Suspension for Subcutaneous Administration (TV-44749) to Oral Olanzapine (European Reference) in Participants With Schizophrenia
Brief Title: An Open-Label Trial to Assess the Comparative Bioavailability of TV-44749 to Oral Olanzapine in Participants With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TV44749-BA-10196; 2023-505664-11-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral olanzapine (Active Comparator)
  Interventions: Drug: Oral olanzapine
- TV-44749 (Experimental)
  Interventions: Drug: TV-44749

INTERVENTIONS:
Drug: TV-44749 — Administered subcutaneously (sc)
  Other Names: Olanzapine
  Arms: TV-44749
Drug: Oral olanzapine — Administered orally
  Other Names: ZYPREXA®
  Arms: Oral olanzapine

SUMMARY:
The primary objective of the study is to evaluate the comparative bioavailability of TV-44749 administered subcutaneous (sc) to oral olanzapine (ZYPREXA®) at steady state in participants with schizophrenia.

A secondary objective of this trial is to evaluate the safety and tolerability of multiple doses of TV-44749 administered sc in participants with schizophrenia.

Another secondary objective of this trial is to compare additional pharmacokinetic parameters of TV-44749 administered sc with oral olanzapine (ZYPREXA®) at steady state in participants with schizophrenia.

The total duration of participation in the trial for each participant is planned to be approximately 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Agree to maintain current smoking or nonsmoking status at the time informed consent is obtained and throughout the trial until completion of the EOT or ET visit (ie, nonsmoking participants must agree not to start smoking and participants who smoke will be excluded if they plan to discontinue smoking during the trial period).
* Have a current confirmed diagnosis of schizophrenia according to an evaluation by the Investigator, as defined by the DSM-5 (American Psychiatric Association 2013a).
* Are clinically stable on oral olanzapine 20 mg daily (ie, dose has not changed in the last 4 weeks) and not currently on other antipsychotic treatments at the time of screening. Participants on alternative olanzapine regimens (eg, 10 mg twice daily) may be considered for inclusion in the trial based upon the Investigator's clinical judgment.
* Women may be included only if they have a negative serum beta human chorionic gonadotropin (HCG) test result at screening; they are surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal (postmenopausal status will be confirmed by a follicle-stimulating hormone screen according to the clinical laboratory standard value) for at least 1 year; or they are practicing a highly effective method of birth control and not planning pregnancy for at least 30 days before the trial, for the duration of the trial, and for 70 days after the last dose administration, if they are sexually active and of childbearing potential.
* Men must be sterile; or if they are potentially of reproductive competence and have sexual relationship with female partners of childbearing potential, they must use, together with their female partners, highly effective birth control methods for the duration of the trial and for 70 days after the last dose administration.

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* History or known risk of narrow-angle glaucoma.
* History or a complication of diabetes (hemoglobin A1c 6.5% or above and/or fasting plasma glucose 126 mg/dL or above).
* Evidence of significant hepatic disorder.
* The participant is a pregnant or lactating woman or plans to become pregnant during the trial or within 70 days after the last dose administration.
* Known hypersensitivity or idiosyncratic reaction to olanzapine (or unable to tolerate oral olanzapine dose) or any of the excipients of TV-44749 in any formulation, their related compounds, or to any metabolites, or any compound listed as being present in TV-44749 or oral olanzapine.
* Presence of excessive pigment, bruises, scars, or tattoos around the potential injection area.
* Personal or family history of arrhythmia, sudden unexplained death at a young age (before 40 years) in a first-degree relative, long QT syndrome, personal history of syncope, or history of uncontrolled high blood pressure. Participants with history of high blood pressure who no longer require treatment or participants who are treated with antihypertensive medications and whose blood pressure is currently well-controlled, may be enrolled.
* Substance use disorder criteria for alcohol, drug, or any other substance dependence (with the exception of nicotine or caffeine) have been met within the past 12 months prior to screening as defined by the DSM-5 (American Psychiatric Association 2013b).
* A current clinically significant DSM-5 diagnosis other than schizophrenia.

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of TV-44749 | Days 57 to 85
AUC of oral olanzapine | 24-hour period following administration of the 7th dose

SECONDARY OUTCOMES:
Number of participants with at least one treatment-emergent adverse event during treatment with TV-44749 | Days 1 to 113
Number of participants with at least one treatment-emergent serious adverse event during treatment with TV-44749 | Days 1 to 113
Number of participants with at least one injection site adverse event during treatment with TV-44749 | Days 1 to 113
Maximum observed plasma drug concentration at steady state (Cmax,ss) of TV-44749 | Day 57 to Day 85
Plasma concentration at the end of the dosing interval at steady state (Ctrough,ss) of TV-44749 | Day 85
Cmax,ss of oral olanzapine | 24-hour period following administration of the 7th dose
Ctrough,ss of oral olanzapine | 24-hour period following administration of the 7th dose

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (9):
- United States (6):
  - Teva Investigational Site 15739, Los Alamitos, California
  - Teva Investigational Site 15740, Torrance, California
  - Teva Investigational Site 15738, Hollywood, Florida
  - Teva Investigational Site 15741, Atlanta, Georgia
  - Teva Investigational Site 15742, Decatur, Georgia
  - Teva Investigational Site 15737, Marlton, New Jersey
- Teva Investigational Site 60053, Zagreb, Croatia
- Teva Investigational Site 31326, Zamora, Spain
- Teva Investigational Site 34310, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.